CLINICAL TRIAL: NCT00765063
Title: A 6 Month, Prospective, Open-Label Multiple Center Extension Trial To Evaluate The Long Term Safety And Sustained Efficacy Of Fragmin In The Treatment Of Chronic Foot Ulcers In Diabetic Patients With Peripheral Arterial Occlusive Disease
Brief Title: The Effect Of Fragmin In The Treatment Of Neuroischaemic Foot Ulcers In Diabetic Patients (A6301086)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A6301086
Record Dates: First submitted 2008-09-30; First posted 2008-10-02 (Estimated); Results first posted 2012-01-13 (Estimated); Last update posted 2012-01-13 (Estimated); Status verified 2011-12

CONDITIONS: Diabetic Foot Ulcer
Keywords: Diabetic Foot Ulcers Neuroischaemic
MeSH Terms: conditions — Diabetic Foot | interventions — Dalteparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Active (Experimental): Active study treatment
  Interventions: Drug: Fragmin

INTERVENTIONS:
Drug: Fragmin — Pre-filled syringes containing a single dose of 5000 IU Fragmin/ Dalteparin Sodium
  Other Names: Dalteparin sodium

SUMMARY:
The primary objective of this 6 month open-label extension trial is to evaluate long-term safety and tolerability of dalteparin in treatment of chronic neuroischaemic foot ulcers in diabetic patients with peripheral arterial occlusive disease (PAOD) and peripheral neuropathy.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have completed the 6 month study duration in the A6301083 study.
* Subjects must have a positive ulcer treatment response, defined as a reduction in the study ulcer area size (ie, ulcer area reduction >0%) at Visit 8 (EOT Visit) from baseline in the A6301083 study.
* All ulcers must have an ulcer staging of 1C, 2C, 1D or 2D according to the University of Texas wound classification system

Exclusion Criteria:

* Subjects who have the following:
* Intact skin healing (defined as 100% reduction in ulcer surface area with full epithelialisation at or prior to the EOT visit in the A6301083 study).
* A study ulcer area at Visit 8 (EOT visit) which is greater or equal to the baseline ulcer area (ie, ulcer area increase ≥0%) in the A6301083 study.
* Subjects with an ulcer grading of 0 or 3 or staging of A or B according to the University of Texas wound classification system.
* Subjects with a known bleeding disorder or evidence of active bleeding.
* Subjects who are on dialysis.
* Subjects who where found to be major protocol violators in A6301083 study.
* Subjects who did not complete the 6 month study period of the A6301083 study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2008-10; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (24):
- Pfizer Investigational Site, Vienna, Austria
- Pfizer Investigational Site, Ransart, Belgium
- Pfizer Investigational Site, Winnipeg, Manitoba, Canada
- Czechia (2):
  - Pfizer Investigational Site, Prague
  - Pfizer Investigational Site, Zlín
- Pfizer Investigational Site, Aarhus C, Denmark
- Pfizer Investigational Site, Karlsbad, Germany
- Pfizer Investigational Site, Melissia/Athens, Greece
- Pfizer Investigational Site, Florence, Italy
- Pfizer Investigational Site, Tønsberg, Norway
- Poland (4):
  - Pfizer Investigational Site, Lodz
  - Pfizer Investigational Site, Puławy
  - Pfizer Investigational Site, Warsaw
  - Pfizer Investigational Site, Wroclaw
- Russia (3):
  - Pfizer Investigational Site, Moscow, Russia
  - Pfizer Investigational Site, Moscow
  - Pfizer Investigational Site, Saint Petersburg
- Sweden (3):
  - Pfizer Investigational Site, Karlstad
  - Pfizer Investigational Site, Malmo
  - Pfizer Investigational Site, Stockholm
- Ukraine (3):
  - Pfizer Investigational Site, Kharkiv
  - Pfizer Investigational Site, Kyiv
  - Pfizer Investigational Site, Lviv
- Pfizer Investigational Site, Birmingham, United Kingdom

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6301086&StudyName=The%20Effect%20Of%20Fragmin%20In%20The%20Treatment%20Of%20Neuroischaemic%20Foot%20Ulcers%20In%20Diabetic%20Patients%20%28A6301086%29

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a follow-up study of A6301083 (NCT00662831)
Groups:
- Dalteparin: Dalteparin sodium 5000 International Units (IU) (0.2 mL) administered subcutaneously (s.c.) once daily (OD) for a maximum duration of 24 weeks.
Period: Overall Study
Arm/Group | Dalteparin
Started | 62
Completed | 30
Not Completed | 32
Not completed — Lack of Efficacy | 5
Not completed — Withdrawal by Subject | 1
Not completed — Other | 16
Not completed — Protocol Violation | 6
Not completed — Adverse Event | 4

BASELINE CHARACTERISTICS:
Arm/Group | Dalteparin
Number analyzed (Participants) | 62
Age Continuous [Mean (Standard Deviation); unit: years] | 65.2 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 46

OUTCOME MEASURES:

1. Primary Outcome: Number of All Hemorrhages
Description: Major hemorrhages: defined as fatal bleeding, clinically overt bleeding causing a fall in hemoglobin greater than or equal to 20 gram (g)/litre (L) (2 g/ decilitre [dL]), clinically overt bleeding leading to transfusion of greater than or equal to 2 units of whole blood or red cells, or symptomatic bleeding in areas of special concern (intracranial, retroperitoneal, intraocular, intraspinal, pericardial, intramuscular with compartmental syndrome, or intraarticular). Minor hemorrhages: defined as bleeding that did not meet the definition of major bleeding.
Time Frame: Baseline to Week 24 (end of treatment [EOT]) or early termination (ET)
Population: Safety analysis population included all participants who were known to have taken at least one dose of the study medication.
Measure: Number; unit: Hemorrhages
Arm/Group | Dalteparin
Number analyzed (Participants) | 62
Hemorrhages | 3

2. Primary Outcome: Number of Major Hemorrhages
Description: Major hemorrhages: defined as fatal bleeding, clinically overt bleeding causing a fall in hemoglobin greater than or equal to 20 g/L (2 g/dL), clinically overt bleeding leading to transfusion of greater than or equal to 2 units of whole blood or red cells, or symptomatic bleeding in areas of special concern (intracranial, retroperitoneal, intraocular, intraspinal, pericardial, intramuscular with compartmental syndrome, or intraarticular).
Time Frame: Baseline to Week 24 (EOT) or ET
Population: as for outcome 1
Measure: Number; unit: Hemorrhages
Arm/Group | Dalteparin
Number analyzed (Participants) | 62
Hemorrhages | 0

3. Primary Outcome: Number of Minor Hemorrhages
Description: Minor hemorrhages: defined as bleeding that did not meet the definition of major bleeding.
Time Frame: Baseline to Week 24 (EOT) or ET
Population: as for outcome 1
Measure: Number; unit: Hemorrhages
Arm/Group | Dalteparin
Number analyzed (Participants) | 62
Hemorrhages | 3

4. Primary Outcome: Number of Clinically Relevant Minor Hemorrhages
Description: Clinically relevant minor (non-major) bleeding was defined as any bleeding compromising hemodynamics, leading to hospitalization, subcutaneous haematoma more than 25 cm^2, intramuscular haematoma, epistaxis lasting for more than 5 minutes, spontaneous gingival bleeding, macroscopic hematuria and gastrointestinal hemorrhage (including at least 1 episode of melaena or hematemesis), rectal blood loss, hemoptysis, and any other bleeding with clinical consequences.
Time Frame: Baseline to Week 24 (EOT) or ET
Population: as for outcome 1
Measure: Number; unit: Hemorrhages
Arm/Group | Dalteparin
Number analyzed (Participants) | 62
Hemorrhages | 2

5. Primary Outcome: Number of Trivial Hemorrhages
Description: Trivial bleeding was defined as all minor bleeding that did not meet the definition of clinically relevant minor bleeding.
Time Frame: Baseline to Week 24 (EOT) or ET
Population: as for outcome 1
Measure: Number; unit: Hemorrhages
Arm/Group | Dalteparin
Number analyzed (Participants) | 62
Hemorrhages | 1

6. Secondary Outcome: Number of Participants With Intact Skin Healing
Description: Intact skin healing was defined as 100 percent reduction in ulcer surface area with full epithelialisation. The ulcer area was measured in square millimetre (mm) by measuring the longest width and length of the ulcer after debridement. The area was calculated from an acetate tracing. Ulcers were also documented by standardized photographs. The largest ulcer was considered the study ulcer in participants with multiple ulcers.
Time Frame: Baseline through Week 24 (EOT) or ET
Population: Intent to treat (ITT) population included all participants who were enrolled into the study.
Measure: Number; unit: Participants
Arm/Group | Dalteparin
Number analyzed (Participants) | 62
Participants | 19

7. Secondary Outcome: Number of Participants With Improved Ulcer Healing
Description: Improved ulcer healing was defined as greater than or equal to 50 percent reduction in ulcer surface area from baseline of the A6301083 study excluding intact skin healing. The ulcer area was measured in square mm by measuring the longest width and length of the ulcer after debridement. Ulcers were also documented by standardized photographs.
Time Frame: Baseline through Week 24 (EOT) or ET
Population: ITT population included all participants who were enrolled into the study.
Measure: Number; unit: Participants
Arm/Group | Dalteparin
Number analyzed (Participants) | 62
Participants | 25

8. Secondary Outcome: Number of Participants Who Underwent Amputation
Description: A major amputation was defined as above the ankle and was reported as below-the-knee and above-the-knee amputations. A minor amputation was defined as below the ankle amputation.
Time Frame: Baseline through Week 24 (EOT) or ET
Population: ITT population included all participants who were enrolled into the study.
Measure: Number; unit: Participants
Arm/Group | Dalteparin
Number analyzed (Participants) | 62
Participants
  All amputations (major and minor) | 1
  Major Amputation | 1
  Minor Amputation | 0

9. Secondary Outcome: Time to Intact Skin Healing
Description: Median time (in months) taken to achieve intact skin healing which was defined as 100 percent reduction in ulcer surface area with full epithelialisation.
Time Frame: Baseline through Week 24 (EOT) or ET
Population: The data was not analyzed as planned because the study enrollment was terminated before the planned number of randomized participants was obtained.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Dalteparin
Number analyzed (Participants) | 0

10. Secondary Outcome: Time to First Amputation
Time Frame: Baseline through Week 24 (EOT) or ET
Population: as for outcome 9
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Dalteparin
Number analyzed (Participants) | 0

11. Secondary Outcome: Number of Participants With Major Cardiovascular Disease Events (MCVE)
Description: MCVE were defined as death due to vascular cause; non-fatal myocardial infarction (MI) excluding procedure related to MI; coronary revascularization procedures not related to MIs; hospitalization for unstable angina or non-fatal stroke.
Time Frame: Baseline through Week 24 (EOT) or ET
Population: as for outcome 9
Measure: Number; unit: Participants
Arm/Group | Dalteparin
Number analyzed (Participants) | 0

12. Secondary Outcome: 11-point Likert Pain Scale
Description: The 11 point Likert pain scale which used a 0 (no pain) to 10 (worst possible pain) point rating system was used to assess participant's pain score. No distinction was made between neuropathy and inflammatory (nociceptive) pain.
Time Frame: Baseline and Week 24 (EOT) or ET
Population: ITT population included all participants who were enrolled into the study.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Dalteparin
Number analyzed (Participants) | 62
Units on a scale
  Baseline | 2.4 (2.1)
  EOT | 2.2 (2.1)

13. Secondary Outcome: 36-Item Short-Form Health Survey (SF-36) Score
Description: SF-36 is a standardized survey evaluating 8 aspects of functional health and well being: physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, mental health. The score for a section is an average of the individual question scores, which are scaled 0-100 (100=highest level of functioning).
Time Frame: Baseline and Week 24 (EOT) or ET
Population: ITT population included all participants who were enrolled into the study. This was calculated only when more than half of the questions within dimension were answered. The 'n' is signifying those participants who received study drug and were evaluated for this measure at the timepoint for each group respectively.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Dalteparin
Number analyzed (Participants) | 62
Units on a scale
  Baseline: Physical Functioning (n= 43) | 34.7 (11.7)
  Baseline: Role-Physical (n= 43) | 36.5 (10.7)
  Baseline: Bodily Pain (n= 43) | 45.1 (9.6)
  Baseline: General Health (n= 43) | 44.1 (4.5)
  Baseline: Visibility (n= 43) | 48.1 (5.7)
  Baseline: Social Functioning (n= 43) | 34.3 (7.6)
  Baseline: Role-Emotional (n= 43) | 36.6 (13.8)
  Baseline: Mental Health (n= 43) | 42.1 (6.4)
  Baseline: Physical (PCS) (n= 43) | 40.1 (7.7)
  Baseline: Mental (MCS) (n= 43) | 41.4 (7.2)
  EOT: Physical Functioning (n= 57) | 34.8 (11.2)
  EOT: Role-Physical (n= 57) | 35.1 (11.0)
  EOT: Bodily Pain (n= 57) | 45.5 (11.3)
  EOT: General Health (n= 57) | 42.9 (4.6)
  EOT: Visibility (n= 57) | 48.7 (6.3)
  EOT: Social Functioning (n= 57) | 35.1 (4.5)
  EOT: Role-Emotional (n= 57) | 36.3 (14.9)
  EOT: Mental Health (n= 57) | 42.2 (7.1)
  EOT: Physical (PCS) (n= 57) | 39.4 (9.0)
  EOT: Mental (MCS) (n= 57) | 41.9 (7.9)

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Dalteparin
Serious Adverse Events (participants affected / at risk) | 11/62
Other Adverse Events (participants affected / at risk) | 26/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dalteparin (N=62)
Anaemia (Blood and lymphatic system disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Cardiac failure acute (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Cellulitis (Infections and infestations) | 2
Erysipelas (Infections and infestations) | 1
Gangrene (Infections and infestations) | 1
Infected skin ulcer (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Carpal tunnel syndrome (Nervous system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dalteparin (N=62)
Anaemia (Blood and lymphatic system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 2
Vertigo (Ear and labyrinth disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Panophthalmitis (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Oedema peripheral (General disorders) | 1
Ulcer haemorrhage (General disorders) | 1
Cystitis (Infections and infestations) | 1
Diabetic foot infection (Infections and infestations) | 3
Erysipelas (Infections and infestations) | 2
Folliculitis (Infections and infestations) | 1
Infected skin ulcer (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 4
Orchitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 1
Tooth infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Wound infection (Infections and infestations) | 1
Chest injury (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 2
Wound (Injury, poisoning and procedural complications) | 1
Body temperature increased (Investigations) | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Osteitis (Musculoskeletal and connective tissue disorders) | 1
Sleep disorder (Psychiatric disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1
Diabetic ulcer (Skin and subcutaneous tissue disorders) | 2
Dry gangrene (Skin and subcutaneous tissue disorders) | 1
Skin discolouration (Skin and subcutaneous tissue disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 4
Urticaria (Skin and subcutaneous tissue disorders) | 1
Tooth extraction (Surgical and medical procedures) | 1
Circulatory collapse (Vascular disorders) | 1
Hypertensive crisis (Vascular disorders) | 1
Intra-abdominal haematoma (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
Study enrollment was terminated before planned number of participants was obtained. Although randomized participants were allowed to complete entire course of therapy according to protocol and study status was therefore designated as completed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.